CLINICAL TRIAL: NCT06124352
Title: Correlation Between Clinical Measurement Scales for Gross Motor Function in Children With Spastic Cerebral Palsy
Brief Title: Correlation Between Clinical Measurement Scales for Gross Motor Function
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Reffat, lecturer at faculty of physical therapy, Cairo University
Other Study IDs: Clinical Measure Scales
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gross Motor Function Measurement - 66 (GMFM- 66) — GMFM-66 was performed for participants established on self-independent motion, with importance on allocations, and motion. The emphasis is to detect the grade that greatest reveals the current skills and disabilities of the child regarding motor functions. The new Gross Motor Ability Estimator (GMAE) scoring method for test-retest reliability data showed a high level of stability of the GMFM-66 over time (ICC=0.9932) that did not differ since the original GMFM 88-item test-retest reliability
Diagnostic Test: Bruininks- Oseretsky Motor Proficiency — The BOT-2 are scale used to evaluate fine and gross motion skill development. It's used to classify children with movement control limitation. The test is appropriate for those aged 4 to 21 years. The interrater reliability ranging from 0.92 to 0.99 and construct validity. r = 0.78 (0.56 - 0.86) (test grades / chronological age)
Diagnostic Test: the Peabody Developmental Motor Scale - Second Edition (PDMS-2 — The PDMS-2 is a consistent test that evaluates a child's movement skills. It is norm-referenced and consists of three composites: Fine Motor (FM), Gross Motor (GM), and Total movement composites (TM). GM composite incorporates 151 points from four sub-tests: reflexes, stationary, locomotion, and object manipulation. A 3-point scale scored for each item, with 2 being the highest score. Definite criterion for score of 2 is given when the child achieves the item, 1 is given when the behavior is emerging but not fully met, and 0 is given when the child cannot achieve the point. The highest raw scores of the sub-tests range from 16 to 198. The test-retest reliability of PDMS-2 was found to be r = 0.85 [24, 25].

SUMMARY:
Evaluating and applying an early and consistent rehabilitation approach to children with neurological impairments requires a multidisciplinary approach that involves different specialists, including pediatricians, pediatric neurologists, professional therapists, and pediatric physical therapists. Evaluation is essential to validate the judgment, monitor the source, and evaluate the mechanical function and related difficulties.

ELIGIBILITY:
Inclusion Criteria:

* children with spastic CP with the capability to keep a standing position alone for at minimum five seconds, and the grade of hypertonicity in the lower extremity varied from grade 1 to grade 2 on the Modified Ashworth Scale with the capability to collaborate and follow directives

Exclusion Criteria:

* Children were excluded If they had a serious neurological condition (epilepsy), orthopedic complications, leg surgery, botulinum toxin treatment in the lower extremity in the last 6 months before the study and suffered from advanced intellectual disability.

Ages: 4 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: In this single-group cross-sectional study design, 50 participants with diplegic CP from the ages of 4 and 6 years evaluated in a physical therapy outpatient clinic and receiving a physiotherapy program for at minimum 6 months were included
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
The principal purpose of this study is to find the correlation between the clinical measurement scales for gross motor function in young CP children | 6 months
  For this study, a correlation between these 3 categories of clinical measures scales was analyzed in diplegic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt